CLINICAL TRIAL: NCT06894355
Title: Group Hydrotherapy Treatment for Athletes With Lower Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gali Dar (Other)
Collaborators: Wingate Institute (Other)
Responsible Party: Sponsor-Investigator, Gali Dar, Prof. Dar , researcher, Department of Physical Therapy, University of Haifa, University of Haifa
Organization: University of Haifa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05/2024
Record Dates: First submitted 2025-01-28; First posted 2025-03-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
Keywords: hydrotherapy, low back pain, group, athlete
MeSH Terms: conditions — Low Back Pain | interventions — Hydrotherapy; Control Groups

STUDY DESIGN:
Intervention Model Description: The interventional group will undergo hydrotherapy treatment in addition to physical therapy treatments The control group will undergo regular physical therapy
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrotherapy (Experimental): Participants will undergo hydrotherapy in addition to regular physical therapy
  Interventions: Other: hydrotherapy
- control (Active Comparator): Participants will go through regular physical therapy treatments

INTERVENTIONS:
Other: hydrotherapy — hydrotherapy in addition to physical therapy
  Arms: Hydrotherapy
Other: control group — regular physical therapy treatments

SUMMARY:
The effect of group hydrotherapy on chronic low back pain and function among athletes will be examined.

DETAILED DESCRIPTION:
Low back pain is a common issue in Western society, especially among athletes who experience significant physical stress. One effective conservative treatment method is hydrotherapy, which involves exercising in water. This approach takes advantage of water's properties, such as buoyancy, weight reduction, and resistance. By using these properties, individuals can perform movements and exercises that may be painful or difficult to do on land.

The purpose of the study is to examine the effect of group hydrotherapy on chronic low back pain and function among athletes.

The study will involve participants with chronic back pain who will complete a 6-week intervention program led by a certified physiotherapist, including hydrotherapy treatment and guidance for independent exercises.

The exercise will include reduced-weight activities at waist-to-neck depth, resistance exercises at varying depths, and the utilization of buoyancy and resistance devices.

The evaluation indicators will be taken before and after the intervention period and will include: a demographic questionnaire, history of back pain and anthropometric details (height, weight), Oswestry questionnaire to assess function following back pain, a visual analog scale to assess the maximum degree of pain during the day, hip range tests, a forward flexion distance test, and a back alignment test. At the end of the intervention, a global rating of scale questionnaire will also be taken to assess the effectiveness of the improvement.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who complain of low back pain for over 3 months,
* VAS>3
* train more than 5 times a week.

Exclusion Criteria:

* acute back pain
* neurological signs (decreased muscle strength, decreased reflexes, radiating to the leg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
change in Visual analog scale | base line, up to 8 weeks
  assessing pain on a scale from 0 (no pain) to 10 (most sever pain). Higher scores means worse outcome.

SECONDARY OUTCOMES:
change in forward flexion distance test | base line, up to 8 weeks
  lumbar flexion assessment by bending forward and measuring distance of fingers from the floor

CONTACTS AND LOCATIONS:
Locations (1):
- Wingate institue, Netanya, Israel

IPD SHARING:
Plan to Share IPD: Yes
outcome measurement results will be shared between therapists performing the study and the principal investigator.
  protocol, results and conclusion will be published via professional paper without patients details.
Supporting Information: Study Protocol, SAP
Time Frame: data will be shared 6 months following the completion of the study
Access Criteria: The principal investigator will share the IPD and supporting information with the therapist performing the intervention.

REFERENCES:
- [Background] Peretro G, Ballico AL, Avelar NC, Haupenthal DPDS, Arcencio L, Haupenthal A. Comparison of aquatic physiotherapy and therapeutic exercise in patients with chronic low back pain. J Bodyw Mov Ther. 2024 Apr;38:399-405. doi: 10.1016/j.jbmt.2023.10.006. Epub 2024 Jan 16. PMID 38763585